CLINICAL TRIAL: NCT03371927
Title: Effect of SINC Feeding Protocol on Weight Gain, Transition to Oral Feeding and the Length of Hospitalization in Premature Infants: Randomized Controlled Study
Brief Title: Effect of SINC Feeding Protocol on Weight Gain, Transition to Oral Feeding and the Length of Hospitalization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Raziye Çelen, Research Assistant, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12.10.2017/34
Record Dates: First submitted 2017-11-30; First posted 2017-12-13 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Feeding; Difficult, Newborn
Keywords: Premature Infants; SINC feeding protocol
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Feeding Method (No Intervention): The control group consisted of prescribed volumes of oral and/or gavage feedings at two or three hour intervals per feeding.
- SINC Feeding Protocol (Experimental): Safe individualized nipple-feeding competence (SINC) protocol
  Interventions: Other: SINC Feeding Protocol

INTERVENTIONS:
Other: SINC Feeding Protocol — Safe individualized nipple-feeding competence protocol for premature infants
  Arms: SINC Feeding Protocol

SUMMARY:
Feeding is one of the most common problems encountered by preterm infants. Besides, effective and safe feeding is one of the important discharge criteria. Feeding problems of premature infants lead to prolonged hospitalization and increased healthcare cost. SINC feeding protocol was developed based on evidence-based feeding protocol (such as cue-based, infant-driven feeding) and individualized developmental care.

The aim of the study is to determine the effect of the SINC feeding protocol on weight gain, transition to oral feeding and the length of hospitalization in premature infants according to traditional feeding method.

Randomized controlled study, including 30 infants of 28-33+6 weeks gestation receiving either Standard Feeding or SINC Feeding Protocol.

ELIGIBILITY:
Inclusion Criteria:

Having been born between 24-33+6 weeks of gestational age 28-33+6 postmenstrual weeks Monitoring with the diagnosis of healthy preterm infants

Exclusion Criteria:

* Receiving mechanical ventilation
* Congenital anomalies
* Having a surgical operation
* Having serious health problems

Ages: 24 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-07-18 (Actual)

PRIMARY OUTCOMES:
Weight Gain | from birth to discharge (average 15 weeks)
  When babies are discharged from the hospital, researchers look at the nursing evolution sheet, their weight gain (gr) along their hospitalization.

SECONDARY OUTCOMES:
Transition to Oral Feeding | from birth to discharge (average 15 weeks)
  time (day) from gavage to full oral feeding

OTHER OUTCOMES:
Length of Hospitalization | from birth to discharge (average 15 weeks)
  When babies are discharged from the hospital, researchers calculate the difference between gestational age (GA) the day they are discharged

CONTACTS AND LOCATIONS:
Overall Officials: Raziye CELEN, PhD, Principal Investigator — Selcuk University; Fatma TAS ARSLAN, Ass.Prof., Study Director — Selcuk Universiy; Hanifi SOYLU, Prof, Study Director — Selcuk University
Locations (1):
- Selcuk University Medical Faculty Hospital, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No